CLINICAL TRIAL: NCT05509829
Title: EvaLuating negAtive pressUre Wound theRapy in brEast coNserving Surgery
Acronym: LAUREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20220056
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Seroma; Wound Complication
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: 150 patients of the prospectively included cohort will undergo NPWT. 150 patients of the retrospective cohort are used as a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPWT group (Experimental): Patients who receive NPWT after surgery.
  Interventions: Device: Negative pressure wound therapy
- Control group (No Intervention): Retrospective cohort who did not receive NPWT.

INTERVENTIONS:
Device: Negative pressure wound therapy — Negative pressure wound therapy using PICO14.
  Arms: NPWT group

SUMMARY:
Negative pressure wound therapy (NPWT) could improve surgical outcomes and reduce complications like SSI, wound dehiscence and seroma in closed surgical wounds. To date, NPWT was not evaluated in patients undergoing breast conserving surgery without direct reconstruction.Therefore, the aim of this trial is to evaluate the feasibility of NPWT after surgery and its effects on postoperative complications.

DETAILED DESCRIPTION:
Rationale:

Negative pressure wound therapy (NPWT) could improve surgical outcomes and reduce complications like SSI, wound dehiscence and seroma in closed surgical wounds. Complication rate after breast conserving surgery for breast cancer is 2-17%, surgical site infections (SSI) being the most common. To date, NPWT was not evaluated in patients undergoing breast conserving surgery without direct reconstruction. Therefore, in this trial, the aim is to evaluate the feasibility of NPWT after breast conserving surgery and its effects on postoperative complications.

Objective and study parameters:

Primary objective is to compare surgical site complications in patients with and without NPWT. Secondary objective is to assess the number of re-interventions, unplanned visits and pain scores.

Study design:

A prospective cohort of 150 patients will be compared to a retrospective cohort of 150 patients.

Study population:

Breast cancer patients undergoing breast conserving surgery with or without sentinel lymph node biopsy.

Intervention (if applicable):

Negative pressure wound therapy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

When participating in this study, patients will need to pay at least one extra visit to the hospital, possibly two if this cannot be combined with the standard postoperative visits. In addition, patients will need to have a device with them for 14 days after surgery. This device is connected to the wound dressing. All wound dressings may cause irritation or an allergic reaction. This risk is not higher than when receiving standard wound dressing, but it is something to take into consideration.

Patients participating in this study may benefit from NPWT regarding the postoperative complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or older.
* Female sex.
* Indication for breast conserving surgery, with or without sentinel lymph node biopsy.

Exclusion Criteria:

* Undergoing mastectomy or modified radical mastectomy.
* Undergoing direct breast reconstruction.
* Patients with a pacemaker, intra cardiac defibrillator (ICD) or other medical device in the proximity of the wound area, due to the magnet in the PICO® device.
* Unable to comprehend implications and extent of the study and/or unable to sign for informed consent.
* Participation in another breast cancer surgery related clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical complications | 3 months after surgery
  Number of surgical complications, including clinically significant seroma, surgical site infections, wound dehiscence or wound necrosis.

SECONDARY OUTCOMES:
Need of re-intervention | 3 months after surgery
  Number of patients who were in need of re-intervention(s) due to the previously mentioned surgical complications
Number of unscheduled visits to the emergency department or outpatient clinic | 3 months after surgery
  Number of unscheduled visits to the emergency department or outpatient clinic
Pain scores during NPWT | one week after surgery
  A numeric rating score will be asked to all patients receiving NPWT.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No